CLINICAL TRIAL: NCT04944108
Title: Does LISA Change the Time of Device Positioning Compared to INSURE in Extremely Low Birth Weight Infants With RDS? A Crossover Randomized Controlled Manikin Trial
Brief Title: LISA vs INSURE in Extremely Low Birth Weight Infants. A Manikin Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOUNIPD
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Distress Syndrome; Preterm Birth; Surfactant Deficiency Syndrome Neonatal
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surfactant administration with less invasive surfactant administration (LISA) approach (Experimental): Participants will be randomized to administer surfactant in a preterm manikin by using the LISA approach (thin catheter)
  Interventions: Procedure: LISA approach
- Surfactant administration with intubation (INSURE) approach (Active Comparator): Participants will be randomized to administer surfactant in a preterm manikin by using the INSURE approach (tracheal tube)
  Interventions: Procedure: Insure approach

INTERVENTIONS:
Procedure: LISA approach — Participants will be randomized to administer surfactant in a preterm manikin by using the LISA approach (thin catheter) or the INSURE approach (tracheal tube)
  Other Names: INSURE approach
  Arms: Surfactant administration with less invasive surfactant administration (LISA) approach
Procedure: Insure approach — Participants will be randomized to administer surfactant in a preterm manikin by using the INSURE approach (tracheal tube)
  Arms: Surfactant administration with intubation (INSURE) approach

SUMMARY:
This is an unblinded, randomized, controlled, crossover (AB/BA) trial of surfactant treatment with LISA vs. INSURE in a manikin simulating an extremely low birth weight infant. Participants will be level III NICU consultants and residents. Randomization will be performed using a computer-generated random assignment list. The primary outcome measure will be the total time of device positioning. The secondary outcomes will be the success of the first and the participant's satisfaction.

DETAILED DESCRIPTION:
Background: Although LISA offers some advantages in ventilation procedure and neonatal outcomes over INSURE, the use of a catheter during LISA may have some drawbacks such as the prolonged duration of the laryngoscopy needed to insert the device. This is likely to aggravate the invasiveness of the procedure, resulting in stressful consequences such as bradycardia, hypoxia and hemodynamic changes.

Objectives: i) time of device positioning, ii) success of the procedure of positioning the device, iii) participant's satisfaction.

Methods: This is an unblinded, randomized, controlled, crossover (AB/BA) trial of surfactant treatment with LISA vs. INSURE in a manikin simulating an extremely low birth weight infant. Participants will be level III NICU consultants and residents. Randomization will be performed using a computer-generated random assignment list. The primary outcome measure will be the total time of device positioning. The secondary outcomes will be the success of the first and the participant's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Level III NICU consultants and residents will be eligible to participate in the study.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Time of device positioning | 10 minutes
  Time needed for the correct positioning of the device into the trachea (thin catheter or tracheal tube). In case of failure, total time will be the sum of time of all attempts.

SECONDARY OUTCOMES:
Success of the procedure at the first attempt | 1 minute
  It refers at the success of the device positioning during the first attempt
Participant's satisfaction | 5 minutes
  At the end of the procedure, all participants will be required to fill a 5-item questionnaire aimed to assess their perception on the procedure (Likert scale)
Number of attempts to insert the device in the trachea | 10 minutes
  It refers to the number of attempts to insert the device in the trachea
Correct depth of the device in the trachea | 10 minutes
  It refers to reaching the correct depth in the trachea as assessed by the external observer using a laryngoscope

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Poliambulanza Breacia, Brescia
  - University Hospital of Padova, Padua

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cavallin F, Bua B, Pasta E, Savio F, Villani PE, Trevisanuto D. Device positioning with LISA vs. INSURE: a crossover randomized controlled manikin trial. J Matern Fetal Neonatal Med. 2022 Dec;35(26):10577-10583. doi: 10.1080/14767058.2022.2134774. Epub 2022 Oct 19. PMID 36261132